CLINICAL TRIAL: NCT03204864
Title: Optimization of Coronary Sinus Lead Placement Targeted to the Longest Right-to-Left Delay
Acronym: Opsite 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michele Brignole (Other)
Responsible Party: Sponsor-Investigator, Michele Brignole, MD, Ospedale del Tigullio, Polo di Lavagna
Organization: Ospedale del Tigullio, Polo di Lavagna (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Ver 5.0
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: HF Patient

STUDY DESIGN:
Intervention Model Description: Phase 1. Conventional CS lead placement
  Phase 2. CS placement guided by RLD measurement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional CS lead placement (Active Comparator): Patients will be implanted with a CRT device with or without defibrillator (P/D) as per standard clinical practice, without CS lead pacing specific optimization.
  Interventions: Device: Conventional CS lead placement
- RLD Group (Experimental): Patients CS placement will be guided by RLD measurement. Physician will place the CS lead in the site of longest RLD with a stable and acceptable pacing threshold.
  Interventions: Device: RLD Group

INTERVENTIONS:
Device: RLD Group — patients CS placement will be guided by RLD measurement. Physician will place the CS lead in the site of longest RLD with a stable and acceptable pacing threshold.
  Other Names: CRT
  Arms: RLD Group
Device: Conventional CS lead placement — Clinical Practice
  Other Names: CRT
  Arms: Conventional CS lead placement

SUMMARY:
This study is a prospective, multi-center, physician-initiated study, with intra-center control arm of patients with advanced heart failure undergoing cardiac resynchronization therapy (CRT) with or without defibrillator therapy.

The purpose of this study is to verify whether optimizing the left ventricular lead position at implantation with the pacing cathode corresponding to the longest RV-to-LV electrical delay may result in a better patient outcome. The RV-to-LV electrical delay will be evaluated with RLD value (ms). RLD is the distance between the Right Ventricular pacing marker (VP) and the maximum peak (or the first maximum peak in case of two equally tall peaks) of the LV bipolar deflection.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, physician-initiated study, with intra-center control arm of patients with advanced heart failure undergoing cardiac resynchronization therapy (CRT) with or without defibrillator therapy.

Approximately 300 patients will be included in the study and followed-up for 6 months. Patients recruitment will consist of two sequential phases:

Phase 1 - Conventional CS lead placement (Conventional subgroup). The first 100 patients will be implanted with a CRT device with or without defibrillator (P/D) as per standard clinical practice, without CS lead pacing specific optimization. In these patients RLD is measured blind to implanting physician who will place CS lead according to his/her clinical practice. Since these patients follow strictly standard clinical practice, their implantation data can be collected prospectively or even retrospectively when available.

Phase 2 - Targeted CS lead placement (RLD subgroup). In the second 200 patients CS placement will be guided by RLD measurement. Physician will place the CS lead in the site of longest RLD with a stable and acceptable pacing threshold.

ELIGIBILITY:
Inclusion Criteria:

* Be in NYHA II or III functional class with approved class I or II standard indications by ESC/EHRA Guidelines
* Either patients in sinus rhythm or in atrial fibrillation. In this latter case patients must perform AV node ablation if complete biventricular stimulation cannot be achieved in >95% of beats
* Patients willing and able to comply with study requirements(patients must indicate their understanding of the study and willingness to participate by signing an appropriate informed consent form)
* Successful LV lead implant

Exclusion Criteria:

* Myocardial Infarction, unstable angina within 40 days prior the enrollment
* Recent cardiac revascularization (PTCA, Stent or CABG) in the 4 weeks prior to enrollment or planned for the 3 months following
* Cerebrovascular Accident (CVA) or Transient Ischemic Attack (TIA) in the 3 months prior the enrollment
* Primary valvular disease
* Unable to comply with the follow up schedule
* Less than 18 years of age
* Pregnant or are planning to become pregnant during the duration of the investigation
* Classification of Status 1 for cardiac transplantation or consideration for transplantation over the next 12 months
* Undergone a cardiac transplantation
* Life expectancy < 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical Composite Score -3 months | 3 months
  Improvement in clinical composite score

SECONDARY OUTCOMES:
Clinical Composite Score-6 months | 6 months
  Clinical composite score evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Michele Brignole, MD, Principal Investigator — Ospedale del Tigullio
Locations (4):
- Italy (4):
  - Ospedale Villa Scassi, Genova
  - Ospedale di Imperia, Imperia
  - Ospedale del Tigullio-Polo di Lavagna, Lavagna
  - Ospedale di Massa, Massa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oddone D, Solari D, Arena G, Mureddu R, Nangah R, Giorgi D, Senatore G, Bottoni N, Giaccardi M, Laffi M, Giammaria M, Sitta N, Marras E, Cipolla E, Di Lorenzo F, Carpi R, Brignole M. Optimization of coronary sinus lead placement targeted to right-to-left delay in patients undergoing cardiac resynchronization therapy. Europace. 2019 Mar 1;21(3):502-510. doi: 10.1093/europace/euy275. PMID 30508076